CLINICAL TRIAL: NCT01684293
Title: Occupational Therapy-Based Cognitive Rehabilitation of Cocaine Abusers: A Pilot Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Collaborators: San Francisco Veterans Affairs Medical Center (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 5K23DA034883-02 (NIH)
Record Dates: First submitted 2012-09-10; First posted 2012-09-12 (Estimated); Last update posted 2019-07-01 (Actual); Status verified 2019-06

CONDITIONS: Mild Cognitive Impairment, So Stated; Cocaine Use Disorder
Keywords: Cocaine; Cognitive Impairment; Cognitive Rehabilitation
MeSH Terms: conditions — Cognitive Dysfunction

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Cognitive Rehabilitation (Experimental): Occupational therapy-based cognitive rehabilitation
  Interventions: Behavioral: Occupational therapy-based cognitive rehabilitation
- Psychoeducation/games (Placebo Comparator): Psychoeducation/games
  Interventions: Behavioral: Psychoeducation/games

INTERVENTIONS:
Behavioral: Occupational therapy-based cognitive rehabilitation — Occupational therapy-based cognitive rehabilitation
  Arms: Cognitive Rehabilitation
Behavioral: Psychoeducation/games — Psychoeducation/games
  Arms: Psychoeducation/games

SUMMARY:
This study integrates a model of occupational-therapy based cognitive rehabilitation as part of a comprehensive treatment plan for cocaine abusers. We hypothesize that cognitive impairment and quality of life would improve and that cocaine use would decrease in those participants receiving occupational-therapy based cognitive rehabilitation.

DETAILED DESCRIPTION:
occupational-therapy based cognitive rehabilitation as part of a comprehensive treatment plan for cocaine abusers

ELIGIBILITY:
Inclusion Criteria:

1. Age 18-65
2. Primary cocaine use disorder (based on DSM-5 criteria) and in at least 3 months of remission
3. At least mild cognitive impairment, defined as = or > 1.5 standard deviations impairment on any 2 performance-based neurocognitive measures
4. Needing to change quality of life, defined as self-identifying at least 2 life areas as needing to change on the Drug User Quality of Life Scale
5. A Veteran at the San Francisco Veterans Affairs Medical Center
6. Currently receiving weekly drug counseling (individual or group; at least 1 hour/week) through an outpatient substance use disorder treatment program

Exclusion Criteria:

1. Inability to speak, read, write, and understand English
2. Inadequate hearing or vision
3. Concurrent substance use disorder (except tobacco or caffeine) not in at least 3 months of remission
4. A psychiatric disorder that will interfere with study participation or will make participation hazardous (e.g., psychosis, suicidal or homicidal ideations, severe anxiety)
5. A depressive disorder classified as severe, defined as a Beck Depression Inventory-II score >29
6. Current diagnosis of a bipolar disorder needing acute inpatient psychiatric hospitalization
7. Currently symptomatic from attention-deficit/hyperactivity disorder (DSM-5 criteria)
8. Any learning disorder, any type of dementia, any type of delirium, or an amnestic disorder due to any general medical condition
9. Wechsler Test of Adult Reading standard score <70
10. Mini-Mental State Examination score <24
11. Current use of scheduled (i.e., prescribed) regular (i.e., daily) psychotropics or other medicines with a high likelihood of sedation & cognitive impairment (e.g., benzodiazepines, clozapine, anticholinergics)
12. Currently prescribed stimulants (e.g., methylphenidate) or cognitive enhancers (e.g., donepezil, memantine)
13. Active medical illnesses - uncontrolled diabetes, uncontrolled hypertension, uncontrolled thyroid dysfunction, or uncontrolled B12/folate deficiency; central nervous system illness with potential cognitive aspects (Parkinson's, or Huntington's dementia); Cirrhosis with complications (e.g., ascites, encephalopathy, jaundice, gastrointestinal bleeding); Needing acute medical hospitalization from HIV sequelae, such as HIV-related opportunistic infection
14. Any history of any type of stroke or brain hemorrhage
15. Any history of traumatic brain injury, intracranial pathology (e.g., tumor), or brain surgery
16. Currently on probation or parole
17. Concurrent participation in another study that medically/administratively interferes with this study

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2013-07; Primary Completion 2019-03-31 (Actual); Study Completion 2019-03-31 (Actual)

PRIMARY OUTCOMES:
Change in cognitive impairment | baseline through 6 months
  Global Deficit Score, range 0 (no impairment) to 5 (severe impairment)

CONTACTS AND LOCATIONS:
Overall Officials: Raj K Kalapatapu, MD, Principal Investigator — University of California, San Francisco
Locations (1):
- University of California, San Francisco & San Francisco Veterans Affairs Medical Center, San Francisco, California, United States